CLINICAL TRIAL: NCT01665469
Title: Effect of Tomato Extracted Lycopene on Postprandial Oxidation and inﬂammation in Healthy
Brief Title: Effect of Tomato Extracted Lycopene on Postprandial Oxidation and inﬂammation in Healthy Weight Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LycoRed Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lyc-2012-02
Record Dates: First submitted 2012-08-09; First posted 2012-08-15 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Postprandial Oxidation and inﬂammation
Keywords: anti oxidation; lycopene; Ox-LDL

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Soft gel capsule without test material
  Interventions: Dietary Supplement: Placebo
- Tomato extracted lycopene (Experimental): Soft gel cups for oral use
  Interventions: Dietary Supplement: Tomato extracted lycopene

INTERVENTIONS:
Dietary Supplement: Tomato extracted lycopene
  Arms: Tomato extracted lycopene
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The hypothesis of the study is that tomato extracted lycopene will be able to decrease postprandial oxidation and inﬂammation in healthy weight men and women when compared to Placebo.

DETAILED DESCRIPTION:
Consumption of a high-fat meal results in a postprandial (fed-state) response characterized by hypertriglyceridemia. Postprandial hypertriglyceridemia increases the oxidation of low-density lipoproteins (LDL) and increases blood concentrations of several biomarkers of inﬂammation. This postprandial lipemia-induced oxidative stress mediated response to a high-fat meal has been suggested as a major contributor to the pathogenesis of atherosclerosis along with other chronic disease states of diabetes and obesity. Consumption of foods rich in antioxidant compounds provides a defence source to compliment endogenous defence systems to protect against oxidative damage during pro-oxidant conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age: 21 - 70 years both inclusive
3. Subject with Body Mass Index: 19- 25 kg/m2 both inclusive
4. Subject with Fasting serum LDL-cholesterol: ≥ 100 mg/dL and < 200 mg/dL
5. Subject with High-sensitivity C-reactive protein (hsCRP) < 1.0 mg/L
6. Subject is willing to take supplement once daily for 4 weeks and undergo other study-related procedures
7. Subject is otherwise is in general good health as determined by the principal investigator
8. Subjects is willing to sign an informed consent form prior to joining the study

Exclusion Criteria:

1. Subjects suffering from overweight defined as BMI > 25 kg/m2
2. Subject that is actively losing weight (e.g. are on a diet) or subjects with greater than 5% change in body weight within 1 month prior to the randomization visit
3. Subject taking lipid-altering drug therapy within six weeks prior to screening. Also excluded are supplements known to have significant lipid altering effects, such as niacin, garlic, omega-3 fatty acids, red yeast rice extract, phytostanols / phytosterols, soluble fiber, chitosan and conjugated linoleic acid
4. Subjects using the following medications: systemic corticosteroids, orlistat, bile acid resins, prescription omega-3 fatty acids, cyclical or non-continuous hormone therapy
5. Subjects that use antioxidant agents or vitamins within 6 weeks prior to inclusion into the study. For subject using vitamin supplementation a 6 week wash out will be required prior to inclusion into the study.
6. Subjects that will not be able to follow dietary proscriptions from the screening visit through the final visit
7. Subjects following any special diet including, but not limited to liquid, high or low protein, raw food, vegetarian or vegan, etc.
8. Subjects with known allergy to tomato, carotenoids, or vitamin E
9. Subjects that smoke (past smokers are allowed if smoking was ceased > 2 years prior to study inclusion)
10. Subjects that has high fasting serum triglyceride
11. Subjects that has a diagnosis of type 1 or type 2 diabetes mellitus
12. Subjects that has high serum thyroid-stimulating hormone
13. Subjects that has aspartate aminotransferase (AST) or alanine transaminase (ALT) > 3 times the upper limit of normal
14. Subjects that has Creatinine ≥ 1.5 mg/dl
15. Subjects that has high-sensitivity C-reactive protein
16. Woman subjects with positive pregnancy test
17. Woman subjects that are breast feeding, pregnant, or planning on becoming pregnant during the duration of the study
18. Subjects with known cardiovascular disease or stroke, except for conditions that are deemed clinically insignificant by Principle Investigator or Sub-investigator, or study site physician (e.g. clinically insignificant atherosclerotic lesions observed by imaging studies).
19. Subject with history of significant gastrointestinal disease such as severe constipation, diarrhea, malabsorptive disease, inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis)
20. Subject with history of severe psychiatric illness which in the opinion of the investigator would interfere with the optimal participation in the study
21. Subject with history of bariatric surgery
22. Subject with history or current use of illegal or "recreational" drugs
23. Subject that used any investigational drug(s) 60 days prior to screening
24. Subject that participate in any other clinical trial while participating in this trial

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Reduction of postprandial Oxidized LDL(OX-LDL) levels following 2 weeks of supplementation with tomato extracted lycopene | Baseline and over 6 hours
  Following two weeks of supplementation the evaluation will be done at baseline,before the high fat meal and during 6 hours following the meal.

SECONDARY OUTCOMES:
Reduction of postprandial triglycerides, glucose, insulin and hsCRP levels following 2 weeks of supplementation with tomato extracted lycopene | Baseline and over 6 hours
  Following two weeks of supplementation the evaluation will be done at baseline,before the high fat meal and during 6 hours following the meal.

OTHER OUTCOMES:
Correlation between the anti-oxidation and anti-inﬂammation effects and serum lycopene, phytofluene and phytoene levels | Baseline and over 6 hours
  Following two weeks of supplementation the evaluation will be done at baseline,before the high fat meal and during 6 hours following the meal.
Number of adverse events recorded during the supplementation period, lycopene compared to placebo | 2 weeks
  safety measurements

CONTACTS AND LOCATIONS:
Overall Officials: David Zeltser, Prof', Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- See also: Data on tomato extracted lycopene — http://www.lycored.com